CLINICAL TRIAL: NCT01254188
Title: Extending Molecular Responses With Nilotinib in Newly Diagnosed Chronic Myeloid Leukemia (CML) Patients in Chronic Phase
Brief Title: Safety and Efficacy of Nilotinib in Newly Diagnosed Chronic Myeloid Leukemia Patients
Acronym: ENESTxtnd
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107E2401; NCT01580059 (obsolete NCT alias)
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia,; CML,; nilotinib,; myelogenous,; Philadelphia chromosome
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome | interventions — nilotinib

ARMS (1):
- Nilotinib (Experimental): 300 mg BID
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — This was an open-label, single-arm, prospective, multi-center, Phase IIIb clinical study with nilotinib 300 mg bid treatment in newly diagnosed CML-CP patients not previously treated with imatinib therapy and diagnosed within 6 months of study entry. For patients insufficiently responding to nilotinib 300 mg bid, the dose may have been increased to 400 mg bid. Among patients with adverse events who had dose reduction, this study also allowed a possible re-escalation to 300 mg bid.
  Other Names: AMN107

SUMMARY:
This study will further investigate the safety and efficacy of nilotinib in newly diagnosed chronic myeloid leukemia patients in the chronic phase

ELIGIBILITY:
Inclusion Criteria:

-Patients with chronic myeloid leukemia in the chronic phase diagnosed within 6 months of study entry

Exclusion Criteria:

* Treatment with tyrosine kinase inhibitor or other antileukemic agents or treatments (including HSCT) for longer than 2 weeks, with exception of hydroxyurea and/or anagrelide
* Uncontrolled congestive heart failure or hypertension
* Myocardial infarction or unstable angina pectoris within past 12 months
* Known T315I mutations
* QTcF >450 msec
* Significant arrhythmias

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2011-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (94):
- Algeria (2):
  - Novartis Investigative Site, Algiers, Bouzareah
  - Novartis Investigative Site, Oran
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Paraná, Entre Ríos Province
- Australia (21):
  - Novartis Investigative Site, Canberra, Australian Capital Territory
  - Novartis Investigative Site, Concord NSW, New South Wales
  - Novartis Investigative Site, Gosford, New South Wales
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Douglas, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Wodonga, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Perth, Western Australia
- Brazil (4):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
- Canada (17):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Saint John, New Brunswick
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Weston, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Egypt (4):
  - Novartis Investigative Site, Cairo, Cairo Governorate
  - Novartis Investigative Site, Al Mansurah
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- India (3):
  - Novartis Investigative Site, Tamil Nadu, Chennai
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Vellore, Tamil Nadu
- Israel (3):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Saida
- Malaysia (2):
  - Novartis Investigative Site, Kuala Selangor
  - Novartis Investigative Site, Pulau Pinang
- Mexico (2):
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
  - Novartis Investigative Site, Hermosillo, Sonora
- Novartis Investigative Site, Muscat, Oman
- Russia (13):
  - Novartis Investigative Site, Arkhangelsk, Russia
  - Novartis Investigative Site, Novosibirsk, Russia
  - Novartis Investigative Site, Perm, Russia
  - Novartis Investigative Site, Ryazan, Russia
  - Novartis Investigative Site, Saint Petersburg, Russia
  - Novartis Investigative Site, Tyumen, Russia
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Yekaterinburg
- Saudi Arabia (3):
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh
- South Africa (5):
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Observatory
  - Novartis Investigative Site, Parktown
  - Novartis Investigative Site, Pretoria
- Taiwan (4):
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Linkou District
- Thailand (2):
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Muang
- Tunisia (2):
  - Novartis Investigative Site, Sousse, Tunisie
  - Novartis Investigative Site, Tunis
- Novartis Investigative Site, Dubai, United Arab Emirates

REFERENCES:
- [Derived] Hughes TP, Munhoz E, Aurelio Salvino M, Ong TC, Elhaddad A, Shortt J, Quach H, Pavlovsky C, Louw VJ, Shih LY, Turkina AG, Meillon L, Jin Y, Acharya S, Dalal D, Lipton JH. Nilotinib dose-optimization in newly diagnosed chronic myeloid leukaemia in chronic phase: final results from ENESTxtnd. Br J Haematol. 2017 Oct;179(2):219-228. doi: 10.1111/bjh.14829. Epub 2017 Jul 12. PMID 28699641

RESULTS

PARTICIPANT FLOW:
Groups:
- Nilotinib: Nilotinib 300 mg BID
Period: Overall Study
Arm/Group | Nilotinib
Started | 421
Completed | 328
Not Completed | 93
Not completed — Disease Progression | 6
Not completed — Protocol Violation | 6
Not completed — Pregnancy | 2
Not completed — Death | 4
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 43
Not completed — per investigator discretion | 20

BASELINE CHARACTERISTICS:
Population: Newly diagnosed CML-CP patients not previously treated with imatinib and diagnosed within 6 months of study entry, except for hydroxyurea, and/or anagrelide . In emergent cases where the patient requires disease management Gleevec/Glivec at any dose may be prescribed to the patient for no longer than 2 weeks in duration
Arm/Group | Nilotinib
Number analyzed (Participants) | 421
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 368
  >=65 years | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.13 (14.892)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195
  Male | 226

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Achieving MMR by 12 Months
Description: MMR is defined as BCR-ABL ratio (%) on IS <= 0.1% (corresponds to >=3 log reduction of BCR-ABL transcripts from standardized baseline value). Clopper-Pearson method
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 421
percentage of participants | 70.8 [66.1 to 75.2]

2. Secondary Outcome: Time to Molecular Response at 24 Months
Description: Estimated median time to first MMR by Kaplan-Meier method
Time Frame: 24 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib
Number analyzed (Participants) | 421
Months | 6.0 [5.9 to 6.1]

3. Secondary Outcome: Duration of Major Molecular Response
Description: Kaplan-Meier estimates of duration of first MMR among patients who achieved MMR (FAS) Duration of first MMR (months) = (Minimum date of (loss of first MMR , CML-related death, progression to AP/BC during study treatment, censoring) - date of first MMR + 1) / 30.4375
Time Frame: 3, 6, 9, 12, 15, 18, 21, 24 Months after MMR was detected
Population: Full Analysis set, Number of events / censored 29/312.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 421
percentage of participants
  K-M Estimate for 3 Month Duration | 100 [100 to 100]
  K-M Estimate for 6 Month Duration | 97.1 [65.2 to 99.0]
  K-M Estimate for 9 Month Duration | 92.8 [89.9 to 95.7]
  K-M Estimate for 12 Month Duration | 92.1 [89.1 to 95.1]
  K-M Estimate for 15 Month Duration | 91.7 [88.5 to 94.8]
  18 months | 90.8 [87.4 to 94.1]
  K-M Estimate for 21 Month Duration | 89.7 [85.7 to 93.6]
  K-M Estimate for 24 Month Duration | 85.2 [75.8 to 94.5]

4. Secondary Outcome: Complete Cytogenetic Response
Description: Complete cytogenetic response (CCyR) is defined as a value of 0% Ph+ metaphases in bone marrow.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 421
percentage of participants | 58.7 [53.8 to 63.4]

5. Secondary Outcome: Percentage of Participants Estimated to Maintain Their First CCyR for 6, 12, 18, and 24 Months After the First CCyR Was Achieved as Determined by Kaplan Meier Estimatation.
Description: * CCyR = 0% Ph+ metaphases based on at least 20 metaphases from bone marrow cytogenetics.
  Duration of first CCyR (months) = (date of CCyR loss or censoring - date of first CCyR +1) / 30.4375
Time Frame: 6,12,18 and 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 421
percentage of participants
  6 mos after the first CCyR was achieved | 100 [100 to 100]
  12 mos after the first CCyR was achieved | 99.6 [98.8 to 100]
  18 mos after the first CCyR was achieved | 98.7 [97.1 to 100]
  24 mos after the first CCyR was achieved | 98.7 [97.1 to 100]

6. Secondary Outcome: Overall Survival
Description: OS was defined as the time between date of study entry and date of death due to any cause at any time during the study, including the follow-up period after discontinuation of treatment.
Time Frame: 3, 6, 9, 12, 15, 18, 21, 24 Months
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Nilotinib
Number analyzed (Participants) | 421
percentage probability
  3 months K-M Estimate | 99.8 [99.3 to 100]
  6 months K-M Estimate | 99.5 [98.9 to 100]
  9 months K-M Estimate | 99.5 [98.9 to 100]
  12 months K-M Estimate | 99.0 [98.0 to 100]
  15 months K-M Estimate | 98.2 [96.9 to 99.5]
  18 months K-M Estimate | 97.6 [96.1 to 99.2]
  21 months K-M Estimate | 97.6 [96.1 to 99.2]
  24 months K-M Estimate | 97.6 [96.1 to 99.2]

7. Secondary Outcome: Kaplan-Meier Estimates of Progression-free Survival
Description: PFS was defined as the time from the date of study entry to the date of event defined as the first documented disease progression to AP/BC or the date of death from any cause occurring on treatment.
Time Frame: 3,6,9,12,15,18,21,and 24 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Nilotinib
Number analyzed (Participants) | 421
percentage probability
  3 mos | 99.7 [99.3 to 100]
  6 mos | 99.5 [98.8 to 100]
  9 mos | 98.9 [97.8 to 100]
  12 mos | 98.6 [97.4 to 99.8]
  15 mos | 98.0 [96.5 to 99.5]
  18 mos | 97.6 [96.0 to 99.3]
  21 mos | 97.6 [96.0 to 99.3]
  24 mos | 97.0 [95.1 to 98.8]

8. Secondary Outcome: Kaplan-Meier Estimates of Failure-free Survival
Description: Time to event (months) = (date of event or censoring - date of study entry + 1) / 30.4375. Date of event is the earliest date of the following events during treatment : discontinuation of nilotinib for nilotinib-related adverse events, death due to any cause, progression to AP or BC, loss of PCyR, loss of CCyR, loss of CHR. Time is censored at the date of last assessment in the trial for patients without event.
Time Frame: 3,6,9,12,15,18,21,and 24 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Nilotinib
Number analyzed (Participants) | 421
percentage probability
  3 mos | 97.4 [95.8 to 98.9]
  6 mos | 95.9 [93.9 to 97.8]
  9 mos | 94.6 [92.4 to 96.8]
  12 mos | 93.6 [91.2 to 96.0]
  15 mos | 92.0 [89.4 to 94.7]
  18 mos | 91.0 [88.2 to 93.8]
  21 mos | 89.7 [86.6 to 92.7]
  24 mos | 88.8 [85.7 to 92.0]

ADVERSE EVENTS:
Arm/Group | Nilotinib
Serious Adverse Events (participants affected / at risk) | 97/421
Other Adverse Events (participants affected / at risk) | 357/421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=421)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 1
ANAEMIA (Blood and lymphatic system disorders) | 4
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 3
PANCYTOPENIA (Blood and lymphatic system disorders) | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 12
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2
ANGINA PECTORIS (Cardiac disorders) | 2
ANGINA UNSTABLE (Cardiac disorders) | 3
ARRHYTHMIA (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 4
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
CARDIAC TAMPONADE (Cardiac disorders) | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2
SINUS BRADYCARDIA (Cardiac disorders) | 1
HYPERTHYROIDISM (Endocrine disorders) | 1
CATARACT (Eye disorders) | 2
RETINAL VEIN OCCLUSION (Eye disorders) | 1
VITREOUS HAEMORRHAGE (Eye disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 2
DUODENAL ULCER (Gastrointestinal disorders) | 1
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1
INTESTINAL INFARCTION (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 7
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 1
GENERALISED OEDEMA (General disorders) | 1
PAIN (General disorders) | 1
PYREXIA (General disorders) | 3
SUDDEN DEATH (General disorders) | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2
CHOLELITHIASIS (Hepatobiliary disorders) | 1
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1
ANAL ABSCESS (Infections and infestations) | 1
APPENDICITIS (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
DIARRHOEA INFECTIOUS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 4
PYELONEPHRITIS CHRONIC (Infections and infestations) | 1
TRACHEOBRONCHITIS (Infections and infestations) | 1
LACERATION (Injury, poisoning and procedural complications) | 2
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1
AMYLASE INCREASED (Investigations) | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 2
LIPASE INCREASED (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPERLIPASAEMIA (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BLAST CELL CRISIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBRAL HAEMATOMA (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1
MYASTHENIA GRAVIS (Nervous system disorders) | 1
SCIATICA (Nervous system disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 2
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 1
POLYMENORRHOEA (Reproductive system and breast disorders) | 1
PROSTATITIS (Reproductive system and breast disorders) | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
VOCAL CORD CYST (Respiratory, thoracic and mediastinal disorders) | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 2
AORTIC STENOSIS (Vascular disorders) | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=421)
ANAEMIA (Blood and lymphatic system disorders) | 43
NEUTROPENIA (Blood and lymphatic system disorders) | 45
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 78
ABDOMINAL PAIN (Gastrointestinal disorders) | 29
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 30
CONSTIPATION (Gastrointestinal disorders) | 51
DIARRHOEA (Gastrointestinal disorders) | 41
DYSPEPSIA (Gastrointestinal disorders) | 30
NAUSEA (Gastrointestinal disorders) | 60
VOMITING (Gastrointestinal disorders) | 29
FATIGUE (General disorders) | 48
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 32
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 44
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 51
AMYLASE INCREASED (Investigations) | 25
BLOOD BILIRUBIN INCREASED (Investigations) | 39
BLOOD CHOLESTEROL INCREASED (Investigations) | 25
LIPASE INCREASED (Investigations) | 66
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 38
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 28
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 24
BACK PAIN (Musculoskeletal and connective tissue disorders) | 28
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 25
MYALGIA (Musculoskeletal and connective tissue disorders) | 32
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 25
DIZZINESS (Nervous system disorders) | 28
HEADACHE (Nervous system disorders) | 77
COUGH (Respiratory, thoracic and mediastinal disorders) | 24
ALOPECIA (Skin and subcutaneous tissue disorders) | 50
DRY SKIN (Skin and subcutaneous tissue disorders) | 28
PRURITUS (Skin and subcutaneous tissue disorders) | 50
RASH (Skin and subcutaneous tissue disorders) | 76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.